CLINICAL TRIAL: NCT00337688
Title: Joystick Use for Virtual Electric Power Wheelchair Driving in Individuals With Spastic Cerebral Palsy
Brief Title: Power Wheelchair Joystick Use in Spastic Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: University of Pittsburgh (Other)
Collaborators: Human Engineering Research Laboratories (Other)
Responsible Party: Sponsor
Other Study IDs: 0512006
Record Dates: First submitted 2006-06-14; First posted 2006-06-16 (Estimated); Last update posted 2011-09-14 (Estimated); Status verified 2011-09

CONDITIONS: Cerebral Palsy; Spasticity
Keywords: Cerebral Palsy; Spasticity; Joystick; Wheelchair; rehabilitation
MeSH Terms: conditions — Cerebral Palsy; Muscle Spasticity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: isometric joystick — isometric joystick

SUMMARY:
There are over 750,000 individuals in the U.S. with Cerebral Palsy (CP). Up to 46% of adults with CP report limited mobility in their communities. However, upper limb spasticity and problems with movement can make the independent use of a wheelchair difficult. Forty percent of individuals who desire mobility via electric wheelchairs are precluded from using them because of problems with upper limb function. No studies to date have produced devices that definitively improve mobility for these individuals. We will recruit 22 subjects with Spastic CP and 22 age and gender matched control subjects without apparent disability from advertisements, mailings, and outpatient clinics. Both a conventional joystick (MSJ) and a novel joystick that is customized for each subject will each be used six different computer screen tasks that simulate driving a wheelchair on a path. We will compare subjects and joysticks based on driving performance. Understanding problems with driving will help us to design joysticks and other assistive devices, not only for CP but for Traumatic Brain Injury, Spinal Cord Injury, Parkinson's Disease, stroke, or a variety of other disabilities.

DETAILED DESCRIPTION:
There are over 750,000 individuals in the U.S. with Cerebral Palsy (CP). Up to 46% of adults with CP report limited mobility in their communities. However, upper limb spasticity and motor control impairment can make the independent use of a wheelchair difficult. Forty percent of individuals who desire mobility via electric wheelchairs are precluded from using them because of problems with upper limb function including motor, sensory, or cognitive impairments that can make the use of a conventional joystick difficult. No studies to date have produced devices that definitively improve mobility for these individuals. We will recruit 22 subjects with Spastic CP and 22 age and gender matched control subjects without apparent disability from advertisements, mailings, and outpatient clinics. Both a conventional motion sensing joystick (MSJ) and a novel isometric joystick that is customized for each subject will each be used to maneuver a sprite on a computer screen in six different tasks. Each task involves a path with 90-degree turns. Two tasks have paths that are completely visible to the subject, while four have paths that appear either immediately or at 1, 2, or 3 seconds ahead of the sprite. Because subjects with CP and control subjects are likely to drive at different speeds, subjects will drive under conditions of freely chosen speed and with speed controlled at 1.2 m/s. Joystick input signals that represent the sprite's velocity and position will be recorded. Changes in direction and speed, average deviation from path center, number of boundary violations, start and stop reaction times, response times to turns, and duration of subject movement will be calculated. We will use a Repeated Measures design, treating speed as a covariate under the condition when it is freely chosen. We hypothesize that, regardless of joystick or speed condition, subjects with Spastic CP will have more direction and speed changes, greater average deviation from path center, more boundary violations, prolonged reaction times and response times to turns, and prolonged subject movement time compared to controls. We hypothesize that, regardless of joystick or speed condition, decreasing warning time before turns will be correlated with more direction and speed changes, greater average deviation from path center, more boundary violations, and prolonged subject movement time and that the magnitude of these changes will be greater for those with Spastic CP. We hypothesize that, regardless of speed condition, subjects with Spastic CP, when using a MSJ compared to the isometric joystick, will have more direction and speed changes, greater average path deviation, more boundary violations, and prolonged subject movement. Understanding driving task deficits and warning time for movement decisions will help to identify customization parameters for joysticks and other assistive devices, not only for CP but for Traumatic Brain Injury, Spinal Cord Injury, Parkinson's Disease, stroke, or a variety of other disabilities.

ELIGIBILITY:
Inclusion criteria:

1. subjects must be between the ages of 12-80
2. subjects must be able to give written informed consent or consent by proxy to participate
3. subjects with the diagnosis of CP must have a score of 2 or 3 on the Modified Ashworth Scale in at least one of the following in the operating limb: wrist flexors, wrist extensors, elbow flexors, or elbow extensors
4. control subjects must have a Modified Ashworth score of 0 for all of the above muscle groups in both upper limbs
5. subjects must have the minimal motor ability necessary to participate in the trial. This will be measured as follows: after 3 trials, subjects must be able to complete a basic virtual driving with an average minimum speed of no less than 1.2 m/s, an average trial time of no more than 18 seconds, and an average deviation of the center of the virtual wheelchair of no more than 1.5 m from the path center, for each of the two joysticks used. These values are derived from Americans with Disabilities Act (ADA) standard dimensions and human walking speed.

Exclusion Criteria:

1. subjects who are not able to tolerate sitting for 2 hours (the estimated length of the experiment)
2. subjects who have active pelvic or thigh wounds (they may be worsened by prolonged sitting)
3. subjects with a history of seizures in the last 90 days (uncontrolled seizures may be induced by a computer screen task)

Ages: 12 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: subjects with CP and controls
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2006-07; Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brad Dicianno, MD, Principal Investigator — Human Engineering Research Laboratories